#### STUDY PROTOCOL

# STUDY ON THE SAFETY OF ADMINISTERING ISONIAZID TO SYSTEMIC LUPUS ERYTHEMATOSUS PATIENTS TO PREVENT TUBERCULOSIS

Unique Protocol ID: IPD-202402.01 Document Date: August 1<sup>st</sup> 2022 NCT Number: N/A



#### Researcher:

Dr. Laniyati Hamijoyo, dr., Sp.PD-KR, M.Kes (8830960018)

Edhyana Sahiratmadja, dr., PhD (0011056602) Bachti Alisjahbana, dr., Sp.PD-KPTI, PhD (8849720016) Guntur Darmawan, dr., Sp.PD

PADJADJARAN UNIVERSITY 2024

#### STUDY PROTOCOL

## STUDY ON THE SAFETY OF ADMINISTERING ISONIAZID TO SYSTEMIC LUPUS ERYTHEMATOSUS PATIENTS TO PREVENT TUBERCULOSIS

#### Researcher:

**Dr. Laniyati Hamijoyo, dr., Sp.PD-KR., M.Kes** - Division of Rheumatology and Immunology, Department of Internal Medicine, Padjajaran University, Hasan Sadikin Hospital Bandung.

**Bachti Alisjahbana, dr, Sp.PD-KPTI, PhD** - Division of Tropical and Infectious Diseases, Department of Internal Medicine, Padjajaran University, Hasan Sadikin Hospital Bandung.

**Edhyana Sahiratmadja, dr., PhD** - Division of Molecular Biology, Department of Biomedical Sciences, Padjajaran University, Hasan Sadikin Hospital Bandung. **Guntur Darmawan, dr., Sp.PD** - Department of Internal Medicine, Krida Wacana Christian University.

#### Aim

This study aims to prove that the administration of Isoniazid (INH) in the prevention of Tuberculosis (TB) in patients with Systemic Lupus Erythematosus (SLE) is safe against liver toxicity and disease recurrence.

#### Research Design

An open-label, randomized, controlled, prospective cohort study evaluating two groups of SLE patients, those receiving INH and pyridoxine for nine months and those not receiving both drugs. Signs and symptoms of drug-induced hepatotoxicity and degree of SLE disease activity were assessed monthly for the first three months (months 1/2, 1, 2, and 3), and then continued every three months for up to one year (months 6, 9, and 12).

#### Introduction

Systemic Lupus Erythematosus (SLE) is a highly complex chronic autoimmune disease that affects multiple organs.<sup>1</sup> The course of the disease is influenced by many things, one of which is infection.<sup>2</sup> SLE patients are more susceptible to infections, due to their disease activity as well as the use of immunosuppressant drugs and glucocorticoids.<sup>3</sup> One of the infections that mainly affects SLE patients is Tuberculosis (TB) infection,<sup>4</sup> especially patients living in Asian areas that are endemic to TB.<sup>5</sup>

TB infection increases the morbidity and mortality of SLE patients, causing more severe disease and death in SLE.<sup>6-17</sup> The World Health Organization (WHO) has established guidelines for TB prevention in HIV patients.<sup>18</sup> Efforts to prevent TB have been made in HIV patients by administering Isoniazid (INH) prophylaxis and found to significantly reduce the incidence of TB in HIV patients by 35%, with good safety data and no significant increase in drug side effects.<sup>19</sup>

Prevention of TB in SLE is controversial, and no guidelines have been issued on the subject. An Indian study found an 82% reduction in the incidence of TB in SLE patients with INH prophylaxis.<sup>20</sup> However, retrospective studies in Hong Kong and Korea found no significant difference between those given and those not given prophylaxis.<sup>13,21</sup> No studies have specifically examined the safety of INH prophylaxis in SLE patients. Research is needed on the safety of INH in SLE patients, especially in terms of toxicity to the liver and its effect on disease recurrence, before further research on its effectiveness in preventing TB in SLE patients.

#### **Research Design and Subjects**

This is a randomized controlled clinical study involving SLE patients at the Rheumatology Polyclinic, Department of Internal Medicine, Padjadjaran University, Hasan Sadikin General Hospital Bandung,

The diagnosis of SLE is based on the 1997 ACR criteria or 2012 SLICC criteria. The screening included *informed consent*, history taking, physical examination, chest X-ray, and laboratory examination (mainly SGOT/SGPT, HBsAg, anti HCV Total). The examination was conducted to ensure that the subjects did not suffer from active TB, and or impaired liver function. Subjects who meet the inclusion criteria will be randomly divided into two groups, the treatment group receiving INH 5 mg/kg/day (maximum 300 mg/day) and pyridoxine 10 mg/day, and the control group receiving neither drug. Routine SLE medications will be continued throughout the study and recorded at each *visit*.

The research design is depicted through the chart below:



#### **Inclusion and Exclusion Criteria**

#### **Inclusion Criteria**

- SLE patients who do not have signs and symptoms of active TB (pulmonary and extrapulmonary),
- SLE patients who are not on TB treatment,
- SLE patients with no history of TB,
- SLE patients who are in remission or low disease activity state (LLDAS), with a history of stable SLE treatment in the last three months and have good liver function,
- Agree to fully participate in this study.

#### **Exclusion Criteria**

- SLE patients who have previous liver dysfunction, including hepatitis B or hepatitis C,
- SLE patients who have a history of allergy to INH,
- SLE patients with malignancy,
- SLE patients who are pregnant.

#### **Variables**

| VARIABLES | DEFINITION | ASSESSMENT | OUTPUTS | DATA TYPE |
|---|---|---|---|---|
| Systemic<br>Lupus<br>Erythematosus<br>(SLE) | ACR 1997 or SLICC<br>2012 criteria <sup>22,23</sup> | History<br>review,<br>physical<br>examination,<br>laboratory<br>examination | Yes/No | Nominal |
| Age | Age at the time of study | History review | Year | Numerical |
| Duration of SLE | Duration from diagnosis of SLE to inclusion in the study. | History review and medical record | Month | Numerical |
| | | confirmation | | |
| Isoniazid (INH)<br>preventive<br>therapy | INH 5 mg/kg/day,<br>max 300 mg/day for<br>nine months | History review | Yes/No | Nominal |
| Tuberculosis | Active TB. | History<br>review,<br>physical<br>examination,<br>Chest X-<br>Ray,<br>and/or<br>AFB/RMT | Yes/No | Nominal |
| | | examination. | | |
| SLE disease<br>activity <sup>25</sup> | Based on the SLE disease activity index (SLEDAI-2K) score: 0 = remission 1-5 = mild 6-11 = moderate | History<br>review,<br>physical<br>examination,<br>laboratory<br>examination | As per score | Nominal |
| | • ≥12 = severe | | | |
| Changes in SLE<br>disease<br>activity <sup>26</sup> | Based on change in SLE disease activity index (SLEDAI-2K) score. Change in score: • increased ≥ 3 = relapse • decreased ≥ 3 = improved • increased but < 3 = active persistent | History<br>review,<br>physical<br>examination,<br>laboratory<br>examination | As per score | Nominal |
| Drug-induced<br>hepatotoxicity<br>(INH) | Increase of more than<br>twice the upper limit of<br>normal SGOT/SGPT<br>values and<br>improvement after<br>drug withdrawal <sup>27</sup> | History<br>review,<br>physical<br>examination,<br>laboratory<br>examination | Yes/No | Nominal |

| R value <sup>28</sup> | Values used to distinguish the type of damage in druginduced hepatotoxicity. R = (SGPT value / upper limit of normal SGPT value) / (ALP value / upper limit of ALP value). | Laboratory<br>examination | As per the result value | Numerical |
|---|---|---|---|---|
| Types of<br>damage in<br>drug-induced<br>hepatotoxicity <sup>28</sup> | Type of damage: • Hepatocellular (SGPT ≥3 upper limit of normal values and R ≥ 5). • Cholestatic (ALP ≥2 upper limit of normal value and R ≤ 2). • Mixed (SGPT ≥3 upper limit of normal, ALP ≥2 upper limit of normal, ALP ≥2 upper limit of normal, and 2 < R < 5). | Laboratory<br>examination | According to the type of damage | Nominal |
| Severity of drug-induced hepatotoxicity <sup>28</sup> | <ul> <li>Grade 0 (No Liver Injury): the patient can tolerate the drugs and there are no signs and symptoms of hepatotoxicity.</li> <li>Grade 1 (Mild Liver Injury): elevated SGPT and/or ALP values, total bilirubin &lt;2.5 upper limit of normal (2.5 mg/dL or 42.75 µmol/L), INR &lt;1.5. Most patients show adaptive processes to liver damage. It may be accompanied or without symptoms, such as fatigue, nausea, anorexia, right upper abdominal pain, jaundice, itching, skin redness, or weight loss.</li> <li>Grade 2 (Moderate Liver Injury): elevated SGPT and/or ALP values,</li> </ul> | History review, physical examination, laboratory examination | As per grade | Ordinal |

with total bilirubin ≥2.5 upper limit of normal or INR ≥1.5. Symptoms and signs of impaired liver function become more apparent.

- Grade 3 (Severe Liver Injury): elevated SGPT and/or ALP, total bilirubin ≥5 upper limit of normal (5 mg/dL or 85.5 µmol/L) with or without INR ≥1.5. Symptoms and signs of hepatic impairment are obvious, indicating the need for hospitalisation. There are no signs and symptoms of hepatic encephalopathy.
- Grade 4 (Acute Liver Failure): evidence of blood clotting disorders with INR ≥1.5 or PTA <40%, signs and symptoms of hepatic encephalopathy, and total bilirubin values ≥10 upper limit of normal (10 mg/dL or 171 µmol/L) or an increase in total bilirubin values ≥1.0 mg/dL (17.1 µmol/L) per day for 26 weeks after the onset of druginduced hepatotoxicity. Patients may develop ascites and other organ dysfunction.
- Grade 5 (Lethal): death caused by drug-induced hepatotoxicity.

| Unexpected events <sup>29</sup> | <ul> <li>Grade 1 Mild; asymptomatic or mild symptoms only; clinical observation or diagnosis only; intervention not indicated.</li> <li>Grade 2 Moderate; minimal, local or non-invasive interventions are indicated; limitation of daily activities based on age.</li> <li>Grade 3 Severe or medically significant, but not life threatening; indication for hospital admission; limitation of independent daily activities.</li> <li>Grade 4 Lifethreatening; indication for rapid/immediate intervention.</li> <li>Grade 5 Lethal; associated with an adverse event.</li> </ul> | History review, physical examination, laboratory examination | As per grade | Ordinal |
|---|---|---|---|---|
| Acid Fast<br>Bacilli (AFB) <sup>30</sup> | Staining technique to<br>see acid fast bacilli<br>(Mycobacterium<br>tuberculosis) from the<br>sample taken | Laboratory<br>examination | Positive/negative | Nominal |
| Rapid<br>Molecular Test<br>(RMT) <sup>31</sup> | Rapid PCR (Polymerase Chain Reaction) testing using the GeneXpert platform that can detect TB bacteria | Laboratory<br>examination | Positive/negative | Nominal |

#### **Research Duration and Time**

This research was conducted from August 2022 to December 2024.

#### Sample size calculation

The sample size calculation was carried out based on INH prophylaxis studies conducted in HIV patients, obtained the risk of *drug reaction* events of RR 1.2, so that with a confidence level of 95%, power 80%, and effect size 0.5, the sample

size of each group was 27 people, plus 10% to 30 people. Thus, the total number of patients involved is 60 people who will be divided into two groups.

#### **Data Analysis**

This study was conducted to assess the safety of INH drug administration in SLE patients by analyzing the increase in SGOT/SGPT values and assessing SLE disease activity measured using SLEDAI. Both will be assessed after two weeks of drug or placebo administration, followed by monthly for the first three months (months 1, 2, 3), then every three months until one year (months 6, 9, 12). Statistical tests used were t-test and/or chi-square by comparing two treatment groups. Results were considered significant when the p value was  $\leq$  0.05. Data processing was performed with SPSS version 26 and Stata version 13.

#### **Outputs**

The incidence of TB in SLE patients, especially in endemic countries, is high at 11.4%<sup>32</sup>. This rate is much higher than the normal population. The administration of isoniazid (INH) has been recommended for TB prophylaxis in HIV patients. However, until now there has no guideline or agreement on the administration of INH as TB prophylaxis in SLE patients. Studies of INH as TB prophylaxis in SLE patients have shown mixed results. Safety is one of the aspects considered, given the risk of drug-induced hepatitis. Therefore, a study to evaluate the safety of TB prophylaxis therapy with INH in SLE patients is very important. Furthermore, this study can serve as a base for further research to evaluate the effectiveness of TB prophylaxis therapy with INH in SLE patients.

#### **Bibliography**

- Yazdany J, Dall'Era M. Definition and classification of lupus and lupus-related disorders. In: Wallace DJ, Hahn BH, editors. DUBOIS' lupus erythematosus and related syndromes. 8th edition. Philadelphia: Elsevier Saunders; 2013. pp. 1-7.
- 2. Lisnevskaia L, Murphy G, Isenberg D. Systemic lupus erythematosus. Lancet 2014; 384:1878-1888.
- 3. Lliopoulos AG, Tsokos GC. Immunopathogenesis and spectrum of infections in systemic lupus erythematosus. Semin ArthritisRheum1996; 25:318-36.
- 4. Jakes RW, Bae SC, Louthrenoo W, Mok CC, Navarra SV, Kwon N. Systematic Review of the Epidemiology of Systemic Lupus Erythematosus in the Asia-Pacific Region: Prevalence, Incidence, Clinical Features, and Mortality. Arthritis Care & Research. 2012; 64 (2): 159-168
- Global tuberculosis report 2020: executive summary. © World Health Organisation 2020. Available at https://apps.who.int/iris/bitstream/handle/10665/337538/9789240016095eng.pdf
- 6. Ahmmed MF, Islam MN, Ferdous S, Azad AK, Ferdous N. Tuberculosis in Systemic Lupus Erythematosus Patients. Mymensingh Med J. 2019 Oct;28(4):797-807. PMID:31599243.
- 7. Hamijoyo L, Candrianita S, Rahmadi AR, Dewi S, Darmawan G, Suryajaya BS, Rainy NR, Hidayat II, Moenardi VN, Wachjudi RG. The clinical characteristics of systemic lupus erythematosus patients in Indonesia: a cohort registry from an Indonesia-based tertiary referral hospital. Lupus. 2019 Nov;28(13):1604-1609. doi: 10.1177/0961203319878499. Epub 2019 Sep 29. PMID: 31566078.
- 8. Tam LS, Li EK, Wong SM, Szeto CC. Risk factors and clinical features for tuberculosis among patients with systemic lupus erythematosus in Hong Kong. Scand J Rheumatol. 2002;31(5):296-300. doi: 10.1080/030097402760375205. PMID: 12455821
- 9. Yun JE, Lee SW, Kim TH, Jun JB, Jung S, Bae SC, Kim TY, Yoo DH. The incidence and clinical characteristics of Mycobacterium tuberculosis infection among systemic lupus erythematosus and rheumatoid arthritis patients in Korea. Clin Exp Rheumatol. 2002 Mar-Apr;20(2):127-32. PMID: 12051389.
- 10. Erdozain JG, Ruiz-Irastorza G, Egurbide MV, Martinez-Berriotxoa A, Aguirre C. High risk of tuberculosis in systemic lupus erythematosus? Lupus. 2006;15(4):232-5. doi: 10.1191/0961203306lu2289xx. PMID: 16686263.
- 11. Sayarlioglu M, Inanc M, Kamali S, Cefle A, Karaman O, Gul A, Ocal L, Aral O, Konice M. Tuberculosis in Turkish patients with systemic lupus erythematosus: increased frequency of extrapulmonary localisation. Lupus. 2004;13(4):274-8. doi: 10.1191/0961203303lu529xx. PMID: 15176665.
- 12. Shyam C, Malaviya AN. Infection-related morbidity in systemic lupus erythematosus: a clinico-epidemiological study from northern India. Rheumatol Int. 1996;16(1):1-3. doi: 10.1007/BF01419946. PMID: 8783414
- 13. Mok MY, Lo Y, Chan TM, Wong WS, Lau CS. Tuberculosis in systemic lupus erythematosus in an endemic area and the role of isoniazid prophylaxis during corticosteroid therapy. J Rheumatol. 2005 Apr;32(4):609-15. PMID: 15801014
- 14. Lao M, Chen D, Wu X, Chen H, Qiu Q, Yang X, Zhan Z. Active tuberculosis in patients with systemic lupus erythematosus from Southern China: a

- retrospective study. Clin Rheumatol. 2019 Feb;38(2):535-543. doi: 10.1007/s10067-018-4303-z. Epub 2018 Sep 23. PMID: 30244432
- 15. Bharath G, Kumar P, Makkar N, Singla P, Soneja M, Biswas A, Wig N. Mortality in systemic lupus erythematosus at a teaching hospital in India: A 5-year retrospective study. J Family Med Prim Care. 2019 Jul;8(7):2511-2515. doi: 10.4103/jfmpc.jfmpc 362 19. PMID: 31463286; PMCID: PMC6691451.
- Pattanaik SS, Muhammed H, Chatterjee R, Naveen R, Lawrence A, Agarwal V, Misra DP, Gupta L, Misra R, Aggarwal A. In-hospital mortality and its predictors in a cohort of SLE from Northern India. Lupus. 2020 Dec;29(14):1971-1977. doi: 10.1177/0961203320961474. Epub 2020 Sep 30. PMID: 32998621.
- 17. Victorio-Navarra ST, Dy EE, Arroyo CG, Torralba TP. Tuberculosis among Filipino patients with systemic lupus erythematosus. Semin Arthritis Rheum. 1996 Dec;26(3):628-34. doi: 10.1016/s0049-0172(96)80013-8. PMID: 8989807
- 18. Guidelines for the Prevention and Treatment of Opportunistic Infections in HIV-Infected Adults and Adolescents: https://aidsinfo.nih.gov/guidelines
- Ayele HT, Mourik MS, Debray TP, Bonten MJ. Isoniazid Prophylactic Therapy for the Prevention of Tuberculosis in HIV Infected Adults: A Systematic Review and Meta-Analysis of Randomised Trials. *PLoS One*. 2015;10(11): e0142290. Published 2015 Nov 9. doi: 10.1371/journal.pone. 0142290.
- 20. Gaitonde S, Pathan E, Sule A, Mittal G, Joshi VR. Efficacy of isoniazid prophylaxis in patients with systemic lupus erythematosus receiving long term steroid treatment. Ann Rheum Dis. 2002 Mar;61(3):251-3. doi: 10.1136/ard.61.3.251. PMID: 11830432; PMCID: PMC1754016
- 21. Moon JY, Kwon HM, Ahn EY, Park JK, Song YW, Lee EB. Efficacy of Isoniazid Chemoprophylaxis in Lupus Nephritis Patients [abstract]. Arthritis Rheumatol. 2015; 67 (suppl 10).(abstract).
- 22. Hochberg MC. Updating the American College of Rheumatology revised criteria for the classification of systemic lupus erythematosus. *Arthritis Rheum*. 1997;40(9):1725.
- 23. Petri M, Orbai AM, Alarcón GS, Gordon C, Merrill JT, Fortin PR, et al. Derivation and validation of the Systemic Lupus International Collaborating Clinics classification criteria for systemic lupus erythematosus. *Arthritis Rheum*. 2012;64(8):2677-86.
- 24. Koesoemadinata RC, McAllister SM, Soetedjo NNM, Ratnaningsih DF, Ruslami R, Kerry S, et. al. Latent TB infection and pulmonary TB disease among patients with diabetes mellitus in Bandung, Indonesia. *Trans. R. Soc. Trop. Med. Hyg.* 2017;111(2): 81-9.
- 25. Polachek A, Gladman AD, Su JD, Urowitz MB. Defining low disease activity in systemic lupus erythematosus. *Arthritis Care Res.* 2017;69(7):997-1003.
- 26. Mikdashi M, Nived O. Measuring disease activity in adults with systemic lupus erythematosus: The challenges of administrative burden and responsiveness to patient concerns in clinical research. *Arthritis Res. Ther.* 2015;17(1):183.
- 27. Benichou C. Criteria for drug-induced liver disorder: Report of an international consensus meeting. *J. Hepatol.* 1990; 11:272-6.
- 28. Yue-cheng Y, Yi-min M, Cheng-wei C, et al. CSH guidelines for the diagnosis and treatment of drug-induced liver injury. Hepatol Int (2017) 11:221-241. DOI 10.1007/s12072-017-9793-2.
- 29. National Cancer Institute. Common terminology criteria for adverse events (CTCAE).

  Available at: <a href="https://ctep.cancer.gov/protocoldevelopment/electronic\_applications/docs/CTCA">https://ctep.cancer.gov/protocoldevelopment/electronic\_applications/docs/CTCA</a>

- E\_v5\_Quick\_Reference\_5x7.pdf. Accessed March 17<sup>th</sup>, 2021.
- 30. Ministry of Health of the Republic of Indonesia. National Guidelines for Medical Services: Tuberculosis Management. Jakarta (2020).
- 31. Blakemore R, Story E, Heib D, Kop J, Banada P, Owen MR, et al. Evaluation of the analytical performance of the Xpert MTB/RIF assay. *Journal of Clinical Microbiology* 2010;48(7):2495-501.
- 32. Hamijoyo L, Candrianita S, Rahmadi AR, Dewi S, Darmawan G, Suryajaya BS, Rainy NR, Hidayat II, Moenardi VN, Wachjudi RG. The clinical characteristics of systemic lupus erythematosus patients in Indonesia: a cohort registry from an Indonesia-based tertiary referral hospital. Lupus. 2019 Nov;28(13):1604-1609. doi: 10.1177/0961203319878499. Epub 2019 Sep 29. PMID: 31566078.

#### Appendix 1

#### **Gantt Chart Timeline Table**

| T 6 A . 11 . 11 | | Year 1 | | | | | | | Year 2 | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Type of Activity | 4 | 5 | 6 | 7 8 | 3 | 9 | 10 | 11 | 12 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 1 | 2 | 3 | 4 |
| Subject Screening | | | | | | | | | | | | | | | | | | | | | | | | | |
| Subject Recruitment | | | | | | | | | | | | | | | | | | | | | | | | | |
| Inspection | | | | | | | | | | | | | | | | | | | | | | | | | |
| Data Analysis | | | | | | | | | | | | | | | | | | | | | | | | | |
| Report Generation | | | | | | | | | | | | | | | | | | | | | | | | | |
| Publication of Results | | | | | | | | | | | | | | | | | | | | | | | | | |

### CRF INH Safety Study in SLE Patients: Initial Screening

| Subject Number MR Number: | Inpatient | | _□ Rheumato | logy Clinic | □F/ <b>M</b> □ | |
|---|---|---|---|---|---|---|
| Date of Birth (da | ny/month/year): | / / | Tel/Phone | :Gender: | LI, III L | |
| Full Address: | | | | | | |
| Occupation: | | Education: | | Ethnic | e: | |
| Marital Status: _ | | oate of SLE diagno | osis ( <i>month/ye</i> | ar): | | |
| | /month/year):// | | | | | |
| Clinical ( | TB, SLE, Liver Disease, I | Pregnancy) | R | outine Lab data screening | g | Chest X-Ray |
| History review | | | Hb | | | |
| | | | Ht | | | |
| | | | Leukocytes | | | |
| | | | Platelets | Basophils | | |
| | | | | Eosinophils | | |
| | | | Count | Neutrophil Rod | | |
| | | | Type | Neutrophil Segment | | |
| | | | -71 | Monocytes | | |
| History: | TD) E 14 D | 1. 77 | | Lymphocytes | | |
| , | TB): □Ever□ Never□ Dor | | ESR | | | |
| | sease: □Ever□ Never□ D | | SGOT | | | |
| 0, | I: □ Yes□ No□ Don't Kno | | SGPT | | | |
| | ncer: □ Yes□ No□ Don't<br>B treatment: □ Yes□ No□ | | HBsAg | | | |
| , | nant□ Yes□ No□ Don't K | | Anti HCV | | | |
| | | LIIOW | Creatinine | | | |
| Physical Examination | on | | | Proteinuria | | |
| | | | Urinalysis | Erythrocytes | | |
| | | | o i i i i i i i i i i i i i i i i i i i | Leukocytes | | |
| | | | | Cylinders | | |
| *When Clinically | y Suspicious of TB | | | | | |
| Date | | Chest X | K-Ray | | AFB | RMT |

Active TB: □ Yes (Clinical/Bacteriological) □ No

#### SLEDAI

| Parameters | Score | Total | Parameters | Score | Total |
|---|---|---|---|---|---|
| Seizures | 8 | | Arthritis | 4 | |
| Psychosis | 8 | | Myositis | 4 | |
| Organic Brain Syndrome | 8 | | Cylinders | 4 | |
| Visual Impairment | 8 | | Haematuria | 4 | |
| Cranial Nerve Abnormalities | 8 | | Proteinuria | 4 | |
| Lupus Headache | 8 | | Piuria | 4 | |
| Cerebrovascular | 8 | | Pleuritis | 2 | |
| Vasculitis | 8 | | Pericarditis | 2 | |
| New Malar Rash | 2 | | Low complement | 2 | |
| Alopecia | 2 | | Anti-dsDNA increased | 2 | |
| New/recurrent ulcers | 2 | | Thrombocytopenia | 1 | |
| Fever | 1 | | Leukopenia | 1 | |

SLEDAI Total Score: \_\_\_\_ □ 0 (Remission) □ 1-5 (Mild) □ 6-11 (Moderate) □≥ 12 (Severe)

**SLE medications:** Take SLE medications regularly: □ Yes □ No

| Medicine | Dosage | Start date | Stop date |
|-------------------------|---------|------------|-----------|
| □ Prednisone/equivalent | mg/day | | |
| □ Pulse Steroids | mg/day | | |
| □ HCQ/CQ | mg/day | | |
| □ Methotrexate | mg/week | | |
| □ Azathioprine | mg/day | | |

| □ MMF | mg/day |
|---------------------|-----------------|
| □ Mycophenolic acid | mg/day |
| □ Leflunomide | mg/day |
| □ Cyclosporin | mg/N |
| □ Tacrolimus | mg/day |
| □ Cyclophosphamide | □NIH□ EuroLupus |
| □ Rituximab | |
| □ More | |

#### CRF INH Safety Study in SLE Patients: Follow Up

| Subject NumberNo Drug Study | | |
|---|---|---|
| Subject Number No Drug Study MR Number: □Inpatient □ Rheumatology Clinic Full Name: Gender: □F/ M □ Date of Birth (day/month/year): / Tel/Phone: | | |
| Pull NameGender. \(\perp \) \(\perp | | |
| Date of Bittii (aay/month/year). | | |
| <u>Visit</u> (months from visit) Date (day/month/year):/ /<br>Take medication regularly: □ Yes□ No | | |
| Clinical | | Laboratory |
| History review | Hb | |
| □ Fever □ Malaise □ Fatigue □ Abdominal Pain □ Nausea | Ht | |
| □ Vomiting□ Icteric | Leukocytes | |
| □ Others: | Platelets | |
| | | Basophils |
| | | Eosinophils |
| | Count | Neut Rod |
| | Type | Neut Segment |
| | | Monocytes |
| | | Lymphocytes |
| | ESR | 7 1 7 |
| Physical Examination | SGOT | |
| | SGPT | |
| | Creatinine | |
| | | Proteinuria |
| | T Tuin - 1i- | Erythrocytes |
| | Urinalysis | Leukocytes |
| | | Cylinders |
| SLEDAI Score: SLEDAI Total Score: □ 0 (Remission) □ 1-5 (Mild) □ 6-11 (Moderate) □≥ 1 SLE Disease Activity: □ Relapse□ Improving□ Persistently Active□ Remission Elevated SGOT/SGPT≥ 2x Upper limit of normal values: □ Yes□ No Liver function disorders: □ Hepatocellular□ Cholestatic□ Mixed Severity: □ 0 (No Liver Injury) □ 1 (Mild Liver Injury) □ 2 (Moderate Liver Injury) □ 3 (Severe Liver Injury) □ 4 (Acute Liver Failure) □ 5 (Lethal) | | |
| Management of Drug-Induced Hepatoxicity | | |
| ☐ INH discontinue ☐ Continue INH Administration ☐ Other medications: | | |
| Drug-induced hepatotoxicity outcomes | | |

## CRF INH Safety Study in SLE Patients: SLE recurrence

| Subject Number Full Name: Data of Birth (day/month/year): | / Tal/Dhana: | Gender: □F/ L □ |
|---|---|---|
| Full Name:Gender: □F/ L □ Date of Birth (day/month/year):/ Tel/Phone: | | |
| <u>Visit</u> (months from visit) D | ate (day/month/year):/_/ | |
| SLEDAI score (at time of screening) | ):□ Remission □ Mild □ Mode | erate Severe |
| Previous SLEDAI scores: | | |
| Diagnosis of SLE Recurrence | | |
| | Clinical (SLE) | |
| Physical Examination | | |
| Management of SLE Recurrence ( ☐ INH discontinue ☐ Continue INH ☐ Changes in SLE medications (see C ☐ Other medications: | RF for SLE medications, any changes | |
| SLE Recurrence Outcome | | |
| Outputs | SLEDAI Score | Date (day/month/year) |
| □ Relapse | | |
| □ Improving | | |
| ☐ Active Persistent | | |
| □ Remission | | |
| □ Died | | |
| □ Others: | | |

## CRF INH Safety Study in SLE Patients: SLE medications

| No Subject Full Name: Date of Birth (day/month/year): / Tel/Phone: | Gender: □F/ M □ |
|---|---|
| <u>Visit</u> ( months from visit) Date (day/month/year):/ / | |
| Take SLE medication regularly: □ Yes □ No | |

#### **SLE** medications

| SLE medications | |
|----------------------------|------------------|
| Medicine | Dosage |
| ☐ Prednisone or equivalent | mg/day |
| □ Pulse Steroids | mg/day |
| □ HCQ/CQ | mg/day |
| ☐ Methotrexate | mg/week |
| ☐ Azathioprine | mg/day |
| □ MMF | mg/day |
| ☐ Mycophenolic acid | mg/day |
| □ Leflunomide | mg/day |
| □ Cyclosporin | mg/N |
| □ Tacrolimus | mg/day |
| □ Cyclophosphamide | □NIH□ Euro Lupus |
| □ Rituximab | |
| □ Belimumab | |
| □ Others: | |

#### **INFORMED CONSENT**

## STUDY ON THE SAFETY OF ADMINISTERING ISONIAZID TO SYSTEMIC LUPUS ERYTHEMATOSUS PATIENTS TO PREVENT TUBERCULOSIS

Unique Protocol ID: IPD-202402.01 Document Date: August 1<sup>st</sup> 2022 NCT Number: N/A



#### Researcher:

Dr. Laniyati Hamijoyo, dr., Sp.PD-KR, M.Kes (8830960018)

Edhyana Sahiratmadja, dr., PhD (0011056602) Bachti Alisjahbana, dr., Sp.PD-KPTI, PhD (8849720016)
Guntur Darmawan, dr., Sp.PD

PADJADJARAN UNIVERSITY

#### **INFORMATION**

## " Study on the Safety of Administering Isoniazid to Systemic Lupus Erythematosus Patients to Prevent Tuberculosis "

I am Dr. Laniyati Hamijoyo, dr., SpPD-KR, I am a rheumatologist at the Faculty of Medicine, Padjadjaran University / Hasan Sadikin Hospital Bandung. My team and I are conducting a study to determine safety of Isoniazid (INH) to prevent Tuberculosis (TB) in Systemic Lupus Erythematosus (SLE) patients. SLE patients are susceptible to TB disease. This is due to their autoimmune condition, as well as the corticosteroid and/or immunosuppressant drugs taken by the patient. Indonesia has the second highest number of TB cases in the world and remains a TB endemic country to date. TB suffered by people with SLE can cause severe problems, especially in terms of disease recurrence (lupus becomes active) which can worsen the patient's condition. Therefore, TB should be prevented. One form of prevention that can be done is the administration of Isoniazid (INH) therapy for nine months. Through this, SLE patients are expected to avoid TB. We invite you to participate in this study. Your participation in this study is voluntary, so you can decide whether or not to participate.

#### **Research Objectives:**

The aim of this study was to determine the safety of Isoniazid (INH) therapy to prevent TB in SLE patients.

#### Why the subject was chosen:

You were selected as a respondent because you met the criteria intended by the researchers, namely SLE patients with a low degree of disease activity/remission, not currently undergoing TB therapy, no history of TB, no symptoms/signs of active TB disease, no liver function disorders, no history of allergy to INH drugs, and willing to participate in this study until completion.

#### **Procedure:**

This study will be conducted by taking blood samples and performing Chest X-Ray for initial screening. If you meet the criteria, you will be divided into two groups. One group will receive INH therapy at a dose of 5 mg/kg BW/day (maximum 300 mg) and vitamin B6 10 mg/day, while the other group will receive placebo (no INH/Vitamin B6). The drugs will be consumed for nine months. The side effects of the drugs and lupus disease activity will be monitored through monthly blood tests in the first three months (months 1/2, 1, 2, 3) and every three months until month 12 (months 6, 9, 12). If necessary, a chest X-Ray and/or sputum examination will be done to confirm whether you have TB or not.

#### Risk and inconvenience:

Possible risks include discomfort during blood collection, hematoma (blue-black bruising) at the site of blood collection and exposure to X-Ray radiation. Other possible risks include nausea, jaundice, bloating, and impaired liver function.

#### Benefits (direct to subject and general):

Public benefit: This study may serve as a guide for physicians treating SLE patients to provide TB preventive therapy, especially for those living in TB-endemic areas.

Direct benefits obtained by the subject: knowing the status of disease activity, getting screened for TB, and obtaining TB prevention therapy.

#### Alternative procedure:

None.

#### Data confidentiality:

We will guarantee the confidentiality of information relating to your identity and will not be known by unauthorized persons. The results of this study will be published without mentioning your identity.

#### Estimated number of subjects to be included:

The subjects to be included in this study were 60 SLE patients.

#### **Volunteerism:**

Your participation in this study is voluntary.

#### **Subject Participation Period:**

This research is planned to take place August 2022 to December 2024. If you have followed the study completely, your participation in this study is considered complete.

#### Subjects may be excluded/resigned from the study:

If during the implementation of the study you want to withdraw or do not want to continue, then you are allowed to withdraw before the data collection process is carried out.

#### Possible financing from health insurance companies or researchers:

No insurance will be provided to you in this study. If side effects occur due to the INH medication, you will be closely monitored and treated for any possible side effects, such as nausea, vomiting or itching. If hospitalization is required, all treatment costs will be the responsibility of the researcher.

#### Incentives and compensation:

If you are willing to participate in this study, you will be compensated in the form of transport money totaling IDR 50,000 per visit (six visits) until the completion of the study.

#### Question:

If there are any questions regarding this study, respondents can contact the researcher at the rheumatology clinic of Dr. Hasan Sadikin Hospital.

#### Researcher:

Dr. Laniyati Hamijo, dr., SpPD-KR Mobile Number: +6281223032863

#### Research Assistant:

dr. Naurah Alzena Hana Dhea Mobile Number: +6281312126312

## APPROVAL AFTER EXPLANATION TO PARTICIPATE IN THE RESEARCH (INFORMED CONSENT)

I have read or obtained an explanation, fully realize, understand, and understand the purpose, benefits, and risks that may arise in the research, and have been given the opportunity to ask questions and have been answered satisfactorily, as well as at any time can withdraw from participation, then I agree / do not agree\*) participate in this study, entitled:

## "Study on the Safety of Administering Isoniazid to Systemic Lupus Erythematosus Patients to Prevent Tuberculosis"

I voluntarily choose to participate in this study without any pressure. I will be given a copy of the explanation sheet and signed consent form for my records.

I agree:

Yes/No \*)

| | Date | Signature (if not possible, thumbprint can be used) |
|---|---|---|
| Participant Name: | | |
| Age: | | |
| Address: | | |
| Researcher Name: | | |
| Witness Name: | | |

<sup>\*)</sup> cross out unnecessary



#### KEMENTERIAN PENDIDIKAN, KEBUDAYAAN, RISET DAN TEKNOLOGI UNIVERSITAS PADJADJARAN KOMISI ETIK PENELITIAN

#### RESEARCH ETHICS COMMITTEE

Jl. Prof. Eyckman No. 38 Bandung 40161 Telp. & Fax. 022-2038697 email: kep@unpad.ac.id, website: kep.unpad.ac.id

No. Reg.: 2110071088

#### PERSETUJUAN ETIK ETHICAL APPROVAL

Nomor: 305/UN6.KEP/EC/2022

Komisi Etik Penelitian Universitas Padjadjaran Bandung, dalam upaya melindungi hak asasi dan kesejahteraan subjek penelitian serta menjamin bahwa penelitian berjalan sesuai dengan pedoman International Conference on Harmonisation - Good Clinical Practice (ICH-GCP) dan aturan lainnya yang berlaku, telah mengkaji dengan teliti dan menyetujui proposal penelitian berjudul:

The Research Ethics Committee Universitas Padjadjaran Bandung, in an effort to protect the basic rights and welfare of the subject of the research and to assure that a research operates in accordance with International Conference on Harmonisation - Good Clinical Practice (ICH-GCP) guidlines and other applicable laws and regulations, has throughly reviewed and approved a reaserch proposal entitled:

"STUDI KEAMANAN PEMBERIAN OBAT ISONIAZID PADA PASIEN LUPUS ERITEMATOSUS SISTEMIK UNTUK MENCEGAH TERJADINYA INFEKSI TUBERKUI OSIS'

Nama Peneliti Utama

Dr. Laniyati Hamijoyo, dr. SpPD-KRM.Kes

Principal Researcher

Pembimbing/Peneliti Lain Supervisor/Other Researcher Edhyana K. Sahiratmadja, dr., Ph.D Bachti Alisjahbana, dr., SpPD-KPTI., PhD

Guntur Dharmawan, dr SpPD

Nama Institusi

Departemen Imunologi Institution

Fakultas Kedokteran Universitas Padjadjaran

proposal tersebut dapat disetujui pelaksanaannya. hereby declare that the proposal is approved.



Ditetapkan di : Bandung

Issued in

Tanggal : 31-03-2022

Date

Ketua, Chairman.

Nur Atik, dr. M.Kes., PhD NIP. 19811010 200801 1 019

#### Keterangan/notes:

Persetujuan etik ini berlaku selama satu tahun sejak tanggal ditetapkan. This ethical clearance is effective for one year from the due date.

Pada akhir penelitian, laporan pelaksanaan penelitian harus diserahkan ke Komisi Etik Penelitian. In the end of the research, progress and final summary report should be submitted to the Research Ethics Committee.

Jika ada perubahan atau penyimpangan protokol dan/atau perpanjangan penelitian, harus mengajukan kembali permohonan kajian etik penelitian. If there be any protocol modification or deviation and/or extension of the study, the Principal Investigator is required to resubmit the protocol for approval. Jika ada kejadian serius yang tidak diinginkan (KTD) harus segera dilaporkan ke Komisi Etik Penelitian.

If there are Serious Adverse Events (SAE) should be immediately reported to the Research Ethics Com